CLINICAL TRIAL: NCT01897220
Title: Perioperative Ischemia Versus Perioperative Bleeding During Non-cardiac Surgery in Cardiac Patients : PRAGUE 14 Study
Brief Title: Perioperative Ischemia Versus Perioperative Bleeding During Non-cardiac Surgery in Cardiac Patients
Acronym: PRAGUE-14
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Principal Investigator, Petr Widimsky, MD, Professor, Charles University, Czech Republic
Other Study IDs: NT/11506-6
Record Dates: First submitted 2013-06-27; First posted 2013-07-11 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Surgical Procedure, Non-cardiac; Cardiovascular Disease Patients; Perioperative Period
Keywords: Noncardiac surgery;; Perioperative ischemic complications;; Perioperative bleeding complications;; Antithrombotic therapy;; Coronary artery disease;; Stent thrombosis;; Perioperative infarction.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- University Hospital Patients: Consecutive patients with cardiovascular disease(s) undergoing non-cardiac surgery

SUMMARY:
The aim of the study is to analyze the present use of antithrombotic therapy on a large cohort of consecutive cardiacs undergoing non-cardiac surgery. If even and for how long the medication was discontinued, if any other antithrombotic therapy was used in the perioperative period and prevalence of perioperative complications - especially ischemic or bleeding. These complications will be correlated with the pattern of antithrombotic therapy administration. Working hypothesis is to obtain a large database of unselected cohort of consecutive patients for mapping of this practically important, but in the evidence-based medicine, still neglected problem.

DETAILED DESCRIPTION:
This project will closely describe (prospective registry) the present situation (anti-thrombotic medication, prevalence of bleeding and ischemic complication) in a large consecutive cohort of non-selected cardiac patients, who are undergoing non-cardiac surgery.

Patients have to meet all three inclusion criteria: (1) Any kind of non-cardiac surgery (acute or elective) performed under general or neuraxial anaesthesia in four surgical departments - General surgery, Orthopedics-Trauma, Urology and Neurosurgery. (2) History of cardiac disease with risk of arterial, intracardiac or vein thrombosis or embolism. (3) Signed Informed consent. All operated patients who meet the inclusion criteria will get enrolled, i.e. all consecutive cardiacs, who signed Informed consent.

Baseline clinical indicators, chronic and perioperative medication, ECG, laboratory tests and all complications (especially ischemic and bleeding) will be registered.

Participants will be followed for the duration of hospital stay, an expected average of 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Any kind of non-cardiac surgery (acute or elective) performed under general or neuraxial anaesthesia in four surgical departments - General surgery, Orthopedics-Trauma, Urology and Neurosurgery.
* History of cardiovascular disease with risk of arterial, intracardiac or vein thrombosis or embolism. (3) Signed Informed consent.

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unselected cohort of consecutive patients undergoing non-cardiac surgery in four surgical clinics of the University Hospital.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of perioperative complications - especially ischemic or bleeding | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Prevalence of perioperative complications - especially ischemic or bleeding; These complications will be correlated with the pattern of antithrombotic therapy administration.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Widimsky, Prof., Principal Investigator — Cardiocentre, Univ. Hospital Královské Vinohrady, Prague, Czech Rep.
Locations (2):
- Czechia (2):
  - Cardiocentre, Univ. Hospital Kralovske Vinohrady, Prague
  - Cardiocentre, Univ. Hospital Královské Vinohrady, Prague

REFERENCES:
- [Derived] Ondrakova M, Motovska Z, Waldauf P, Knot J, Havluj L, Bittner L, Bartoska R, Gurlich R, Krbec M, Dzupa V, Grill R, Widimsky P. Antithrombotic therapy of patients with atrial fibrillation discharged after major non-cardiac surgery. 1-year follow-up. Sub-analysis of PRAGUE 14 study. PLoS One. 2017 May 24;12(5):e0177519. doi: 10.1371/journal.pone.0177519. eCollection 2017. PMID 28542316
- See also: Main manuscript — http://link.springer.com/article/10.1007/s12471-014-0575-3
- See also: Subanalysis — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5443499/